CLINICAL TRIAL: NCT07355075
Title: A Double-Blind, Vehicle-Controlled Study to Assess the Efficacy of GX-03 When Used in a Population of Adult Individuals With Moderate to Severe Eczema
Brief Title: A Study to Assess the Efficacy of GX-03 in Moderate to Severe Eczema (Atopic Dermatitis)
Acronym: GX-03 in AD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Turn Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol/Panel 4604
Record Dates: First submitted 2026-01-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Eczema Atopic Dermatitis; Eczema; Atopic Dermatitis
Keywords: Moderate-Severe AD; Moderate-Severe Eczema; Eczema; Atopic Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: The test article will be distributed to study participants and each participant instructed to use the test article on an area of interest. Each subject will be evaluated using the EASI severity scale, vIGA-AD™ scoring system, and PP-NRS score. Evaluations will occur at baseline and again after 4 and 8 weeks of daily use.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded, vehicle controlled, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GX-03 (Experimental): Treatment Arm
  Interventions: Combination Product: GX-03
- Vehicle (Placebo Comparator): Vehicle Control
  Interventions: Other: Vehicle

INTERVENTIONS:
Combination Product: GX-03 — Topical petrolatum-based ointment
  Arms: GX-03
Other: Vehicle — Ointment carrier
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind, vehicle-controlled clinical study designed to evaluate the efficacy and safety of GX-03, a topically applied emollient, in adult subjects with moderate to severe eczema. Approximately 120 adult participants will be enrolled and randomized in a 1:1 ratio to receive either GX-03 or a petrolatum-based vehicle control for 8 consecutive weeks. Efficacy will be assessed using validated clinical outcome measures, including the Eczema Area and Severity Index (EASI), the Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™), and the Peak Pruritus Numeric Rating Scale (PP-NRS). Safety will be evaluated through monitoring of treatment-emergent adverse events throughout the study period.

DETAILED DESCRIPTION:
This Phase 2, randomized, double-blind, vehicle-controlled study will assess the efficacy and safety of GX-03 in adult individuals aged 18 to 70 years with moderate to severe eczema. Eligible participants will be randomly assigned to receive either GX-03 or a vehicle control, applied topically to affected areas at least twice daily for 8 weeks. The investigational product and vehicle will be identical in appearance and packaging to maintain blinding.

Clinical efficacy will be evaluated at baseline and at Weeks 4 and 8. The primary efficacy endpoint is the change from baseline in Eczema Area and Severity Index (EASI) score at Weeks 4 and 8. Secondary efficacy endpoints include changes from baseline in vIGA-AD™ scores and Peak Pruritus Numeric Rating Scale (PP-NRS) scores at the same time points. Subject-reported outcomes and product preference questionnaires will also be collected as exploratory measures.

Safety assessments will include the collection of spontaneous and solicited adverse events from the first application through the final study visit. Weekly telephone safety check-ins will be conducted during interim weeks, and adverse events will be assessed at all on-site visits. The study is expected to enroll sufficient subjects to ensure that at least 100 participants complete the full 8-week treatment period.

ELIGIBILITY:
Participants must meet all of the following criteria:

* Adults aged 18 to 70 years, inclusive
* Male or female subjects in good general health as determined by medical history
* Presence of visible eczematous skin with disease severity consistent with moderate to severe eczema, as assessed by:
* Eczema Area and Severity Index (EASI) and
* Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™)
* Ability to read, understand, and provide written informed consent in English
* Willingness and ability to comply with study procedures, including study visits and daily topical application
* Agreement to use only the assigned study product on designated areas of interest for the duration of the study

Exclusion Criteria

Individuals meeting any of the following criteria will be excluded:

* Pregnant, breastfeeding, or planning pregnancy during the study
* Presence of any skin condition or dermatologic disease that could interfere with study treatment or assessments
* Use of systemic or topical immunosuppressive therapies, including corticosteroids, within 3 weeks prior to enrollment
* Use of anti-inflammatory medications (e.g., topical steroids, ibuprofen, celecoxib); steroid nasal or ophthalmic drops are permitted
* Use of topical medications at the test sites within 72 hours prior to enrollment
* Damaged or altered skin at or near test sites (e.g., sunburn, tattoos, scars, uneven pigmentation) that could confound evaluations
* Any medical condition that, in the investigator's judgment, places the subject at undue risk or compromises study integrity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity (EASI) | Four and Eight Weeks
  Change in EASI Over 4 and 8 Weeks

SECONDARY OUTCOMES:
Change in Investigator Global Assessment (IGA) | Four and Eight Weeks
  Reduction in Investigator Global Assessment of -2
Change in NRS Max Itch | Four and Eight Weeks
  Change in Patient Itch Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- ALS Global, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Protection of participant privacy and re-identification risks Ongoing regulatory or commercial activities Intellectual property and competitive concerns Resource and practical barriers

REFERENCES:
- See also: Sponsor Website — https://www.turntherapeutics.com